CLINICAL TRIAL: NCT03987204
Title: Ivabradine for Rate Control in Permanent Atrial Fibrillation
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Yale University (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2000022064
Record Dates: First submitted 2019-05-31; First posted 2019-06-14 (Actual); Last update posted 2021-07-02 (Actual); Status verified 2021-06

CONDITIONS: Atrial Fibrillation; Atrial Fibrillation, Persistent
MeSH Terms: conditions — Atrial Fibrillation | interventions — Ivabradine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (1):
- Ivabradine (Experimental): Patients with permanent atrial fibrillation and previously implanted pacemakers who will be started on ivabradine.
  Interventions: Drug: Ivabradine

INTERVENTIONS:
Drug: Ivabradine — Ivabradine will be started and titrated to heart rate slowing of 20 bpm or greater, or an increase in pacing.

SUMMARY:
Ivabradine may be useful as a rate controlling agent in atrial fibrillation without negative effects on hemodynamics and inotropy. The objective in this proof of concept study is to investigate the hypothesis that ivabradine will slow the ventricular response in patients with permanent atrial fibrillation and previously-implanted pacemakers.

DETAILED DESCRIPTION:
In a simple cross-over study, the investigators will evaluate the impact of oral Ivabradine on exercise treadmill test, percent pacing as stored in pacemaker diagnostics, and 6 minute walk test.

Aim/Hypotheses

• To determine if the addition of Ivabradine to baseline cardiac medications slows mean and maximum heart rates in permanent atrial fibrillation

* Ivabradine will lower mean and maximum heart rates on treadmill exercise test, without lowering blood pressure
* Ivabradine will increase percent pacing, and lower rates over time as shown on pacemaker diagnostic data
* Ivabradine will improve exertional symptoms and exercise tolerance due to atrial fibrillation as measured by the Borg's scale during a six-minute walk test.

Study Design

1. Patients with permanent atrial fibrillation will undergo baseline exercise treadmill test, measurement of heart rates and percent pacing from pacemaker diagnostics, and a 6 minute walk test with symptomatic assessment of dyspnea using the Borg's scale score.
2. Oral Ivabradine will be started at 5 mg twice daily, and up-titrated to a maximum dose of 7.5 mg twice daily at 7 days if percent pacing has not increased significantly or rates have not slowed more than 20bpm.
3. Exercise treadmill test, measurement of heart rates and percent pacing from pacemaker diagnostics, and a 6 minute walk test with symptomatic assessment of dyspnea using the Borg's scale score will be repeated at 2 weeks.

ELIGIBILITY:
Inclusion Criteria:

* Patients with stable blood pressures with permanent atrial fibrillation and implanted pacemaker pacing less than 50% of the time, with or without concomitant beta blocker or calcium channel blocker use

Exclusion Criteria:

* Patients with uncontrolled hypertension will be excluded
* To eliminate confounding effects, patients on Digoxin therapy will be excluded
* Patients on anti-arrhythmic therapy
* Patients with pre-excitation on EKG
* Patients who pace > 50% of the time
* Patients with severe Child-Pugh C hepatic impairment

Ages: 21 Years to 90 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 4 (Actual)
Dates: Start 2019-06-15 (Actual); Primary Completion 2019-09-17 (Actual); Study Completion 2019-09-17 (Actual)

PRIMARY OUTCOMES:
Heart Rate in Daily Life | 2 weeks
  Average ventricular heart rate derived using pacemaker interrogation over 2 weeks
Percent Pacing in Daily Life | 2 weeks
  Average percent pacing derived using pacemaker interrogation over 2 weeks
Heart Rate on Treadmill | 2 weeks
  Average ventricular heart rate will be recorded after the patient exercises on a treadmill using a heart rate monitor
Symptoms and Exercise Tolerance | 2 weeks
  Patients will undergo a 6 minute walk test, and symptoms and distance walked as measured by standard 6 minute walk protocol

SECONDARY OUTCOMES:
Blood Pressure | 2 weeks
  Blood pressures will be monitored using a blood pressure cuff with the patient at rest for 10 minutes

CONTACTS AND LOCATIONS:
Overall Officials: Rachel Lampert, MD, Principal Investigator — Yale University; Hyon Jae Lee, MD, Study Director — Yale New Haven Hospital
Locations (1):
- Yale New Haven Hospital, New Haven, Connecticut, United States

IPD SHARING:
Plan to Share IPD: No